CLINICAL TRIAL: NCT06644521
Title: Comparison of Angiogenic Factors in the Placentas of Parturient Women With COVID-19
Brief Title: Angiogenic Factors in the Placentas of Women With COVID-19
Status: Completed | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Other Study IDs: MCBU_Covidplasenta
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: COVID-19; Placenta Diseases; Angiogenesis
Keywords: COVID-19; placenta; VEGF; VEGFR-1; PDGF; immunohistochemistry
MeSH Terms: conditions — COVID-19; Placenta Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Biospecimen Retention: Samples With DNA — placenta tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: COVID-19 group
- Group 2: Control

SUMMARY:
Aim: There have been few studies since the beginning of the pandemic researching the histopathologies and conducting molecular investigations of the placentas of SARS-CoV-2 positive pregnant women. The aim of this study was to analyze the changes in the expression of angiogenic growth factors in the placentas of pregnant women infected with SARS-CoV-2 (the COVID-19 group), and to make comparisons with the placentas of non-infected pregnant women (the control group).

Methods: Placentas taken at birth from 20 healthy women (control) and 20 women with a positive test for COVID-19 were prepared for histopathological examination. Immunohistochemical staining was applied in placental tissues with ACE2 (Angiotensin-conversion enzyme-2), VEGF (Vascular Endothelial Growth Factor), VEGFR-1 (Vascular Endothelial Growth Factor Receptor 1) and PDGF (Platelet-Derived Growth Factor).

Results: First, the presence of COVID-19 in the placental tissue was assessed by the ACE2 immunohistochemical method. It was seen that ACE2 was expressed weakly in the placental syncytiotrophoblast cells of non-infected women, but in the syncytiotrophoblasts of the placentas of women infected with COVID-19, ACE2 expression was much higher. VEGF in the endothelial and stromal cells of the villi of the control group was very strong, but in the villi of infected placentas it was significantly weaker. VEGFR-1 was positive in the endothelial membranes of the villi of the control group, but was significantly weaker in the villi of infected placentas. PDGF expression was strong in the syncytiotrophoblast and stromal cells of the control group, but was significantly noticeably weaker in COVID-19 positive placentas.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 patients while pregnancy
* Age range 18-50
* Being literate in Turkish
* Not having any additional disease
* Agreeing to participate in the study

Exclusion Criteria:

* High-risk pregnancies (gestational hypertension, preeclampsia, HELLP syndrome, chronic hypertension, gestational and pregestational diabetes, cholestasis, intrauterine growth retardation, etc.)
* Multiple pregnancy
* Pregnant women under the age of 18
* Smoking
* Medication use (excluding routinely used food supplements during pregnancy)
* Additional disease (thyroid, renal failure, liver failure, hepatitis, heart disease, connective tissue disease, etc.)
* Immunosuppressive use
* Presence of active or chronic infection
* Presence of active or chronic inflammatory disease
* Patients who gave birth at an external center or later chose to withdraw from the study
* Patients who did not have Covid-19 while pregnancy included in the control group

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Covid-19 patients while pregnancy
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Number of 40 participant include this stuedy. Taken 2% of Covid-19 placenta tissues and 2% of normal placenta tissues while birth. Placenta tissues were stained by ACE2, VEGF, VEGFR-1, PDGF immunohistochemistry. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar University, Manisa, Turkey (Türkiye)